CLINICAL TRIAL: NCT02468817
Title: PTH And Calcium Responses to Exercise (PACE) in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 15-0250
Record Dates: First submitted 2015-06-02; First posted 2015-06-11 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Osteoporosis
Keywords: parathyroid hormone (PTH); bone mineral density (BMD)
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treadmill Exercise (Active Comparator): 2 (two) 1-hour of vigorous exercise bouts under different thermal conditions, one at 16 degrees C and one at 26 degrees C.
  Interventions: Procedure: Treadmill Exercise
- Magnitude of Ca loss during Exercise at 26 degrees Celcius (Experimental): Blood samples at 15-min intervals starting 15 min before exercise and ending 60 min after exercise.
  Interventions: Procedure: Magnitude of Ca loss during Exercise at 26 degrees Celcius

INTERVENTIONS:
Procedure: Treadmill Exercise — 2 (two) 1-hour of vigorous exercise bouts under different thermal conditions
  Arms: Treadmill Exercise
Procedure: Magnitude of Ca loss during Exercise at 26 degrees Celcius — Blood samples at 15-min intervals starting 15 min before exercise and ending 60 min after exercise
  Arms: Magnitude of Ca loss during Exercise at 26 degrees Celcius

SUMMARY:
Exercise that causes a decline in serum Calcium (Ca) as a result of dermal Ca loss stimulates bone resorption via an increase in Parathyroid Hormone (PTH).

DETAILED DESCRIPTION:
Determine whether the magnitude of dermal Ca loss (i.e., sweating) during exercise is a determinant of the decline in iCa and increases in PTH and carboxy-terminal collagen crosslinks (CTX; marker of bone resorption). The proposed experiment will address this by manipulating the rate of dermal Ca loss (moderate vs high sweating rate) to determine whether this is the trigger for the cascade described in Figure 1. This will be achieved by having participants perform two identical exercise bouts under different thermal conditions (warm vs cool).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 60-80 y

Exclusion Criteria:

* Use of medications in the past 6 months known to affect bone metabolism (e.g., bisphosphonates, thiazide diuretics, oral glucocorticoids)
* BMD t score < -2.5 at the total hip or lumbar spine
* Known disease or condition associated with intestinal malabsorption
* Moderate or severe renal impairment defined as an estimated glomerular filtration rate of <60 mL/min/1.73m2 based on the MDRD equation
* Chronic hepatobiliary disease, defined as liver function tests (AST, ALT) >1.5 times the upper limit of normal; if such values are obtained on initial screening and thought to be transient in nature, repeated testing will be allowed
* Thyroid dysfunction, defined as an ultrasensitive TSH <0.5 or >5.0 mU/L; volunteers with abnormal TSH values will be re-considered for participation in the study after follow-up evaluation by the PCP with initiation or adjustment of thyroid hormone replacement
* Serum calcium <8.5 or >10.3 mg/dL
* Serum 25(OH)D <20 ng/mL; volunteers with abnormal serum 25(OH)D values may be re-considered for participation in the study if serum 25(OH)D is >20 ng/mL after vitamin D supplementation
* Uncontrolled hypertension defined as resting systolic BP >150 mmHg or diastolic BP>90 mmHg; participants who do not meet these criteria at first screening will be re-evaluated, including after follow-up evaluation by the PCP with initiation or adjustment of anti-hypertensive medications
* History of type 1 or type 2 diabetes
* Cardiovascular disease; subjective or objective indicators of ischemic heart disease (e.g., angina, ST segment depression) or serious arrhythmias at rest or during the graded exercise test (GXT) without follow-up evaluation will be cause for exclusion; follow-up evaluation must include diagnostic testing (e.g., stress echocardiogram or thallium stress test) with interpretation by a cardiologist
* Diagnosis or history of asthma

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-08; Primary Completion 2017-06 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change in Parathyroid Hormone (PTH) | 60 minutes of exercise and 2 hours of recovery
  PTH will be measured during baseline, throughout exercise, and during recovery at regular intervals. We are looking to see how PTH changes over the course of the exercise and recovery period in both the warm and cool conditions. We anticipate that PTH will be higher in the warm condition versus the cool. We expect that men and women will respond similarly.
Change C-Telopeptide (CTX) | 60 minutes of exercise and 2 hours of recovery
  CTX will be measured during baseline, throughout exercise, and during recovery at regular intervals. We are looking to see how PTH changes over the course of the exercise and recovery period in both the warm and cool conditions. We anticipate that CTX will be higher during exercise and recovery in the warm condition versus the cool.
Change in Serum Ionized Calcium (iCa) | 60 minutes of exercise
  iCa will be measured during baseline, throughout exercise, and during recovery at regular intervals. We are looking to see how PTH changes over the course of the exercise and recovery period in both the warm and cool conditions. We expect that serum iCa will be higher in the cool condition versus the warm.
Change in Total Ca | 60 minutes of exercise
  Total Ca will be measured during baseline, throughout exercise, and during recovery at regular intervals. We are looking to see how PTH changes over the course of the exercise and recovery period in both the warm and cool conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah J Wherry, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States